

## STATISTICAL ANALYSIS PLAN

Protocol Number: 1820202

Title: A Phase 2a, Multicenter, Open-Label, Dose-Escalation Study to Evaluate

the Efficacy and Safety of DaxibotulinumtoxinA (DAXI) for Injection for the Treatment of Dynamic Forehead Lines (Frontalis) Following Glabellar

Line Injections

Study Phase: 2a

Sponsor: Revance Therapeutics, Inc.

7555 Gateway Blvd. Newark, CA 94560

SAP Date: 06 Apr 2020

SAP Version Number: Version 2.0

Protocol Version: 04 March 2019





# TABLE OF CONTENTS

| TA | BLE | OF CO | NTENTS | 4 |
|-----|-------|---------|--------------------------------------------|-----|
| LIS | ST OF | TABL | ES | 7 |
| LIS | ST OF | ABBR | EVIATIONS AND DEFINITIONS OF TERMS | 8 |
| 1. | INT | RODUC | CTION | 9 |
| 2. | STU | JDY OB | BJECTIVES | 9 |
| | 2.1 | Objec | tives | |
| | | 2.1.1 | Primary Objective | 9 |
| | 2.2 | | Endpoints | |
| | | 2.2.1 | Efficacy Endpoints | |
| | | 2.2.2 | Safety Endpoints | |
| 3. | | | STUDY DESIGN AND PLAN | |
| | 3.1 | | Design | |
| | | 3.1.1 | Determination of Sample Size | |
| | 2.0 | 3.1.2 | Treatments Administered. | |
| | 3.2 | | acy and Safety Assessments | |
| | | 3.2.1 | Frown and Forehead Wrinkle Severity | |
| | | 3.2.2 | Patient Global Satisfaction with Treatment | |
| | | 3.2.3 | Global Aesthetic Improvement Scale | 1 / |
| | | 3.2.5 | Facial Age Self Evaluation | 10 |
| | | 3.2.5 | FACE-Q <sup>TM</sup> | |
| | | 3.2.0 | TACL-Q | 18 |
| | 3.3 | Safety | Assessments | 18 |
| | 3.3 | 3.3.1 | Adverse Events | |
| | | 31311 | Travelle Evente | |
| | | 3.3.3 | Injection Site Evaluation | 18 |
| | | 3.3.4 | Clinical Laboratory Data | |
| | | 3.3.6 | Vital Signs | 20 |
| | | 3.3.7 | Physical Examination | 20 |
| | 3.4 | Interir | m Analyses and Data Monitoring | 20 |
| | | 3.4.1 | Data Review Committee | 20 |
| | | 3.4.2 | Interim Analysis | 21 |

| 4. | ANA | ALYSIS | POPULATIONS AND SUMMARY GROUPS | 21 |
|---|---|---|---|---|
| | 4.1 | Enroll | ed Population | 21 |
| | 4.2 | GL-Ev | valuable Population | 21 |
| | 4.3 | FHL-E | Evaluable Population | 21 |
| | 4.4 | Safety | Population | 21 |
| | 4.5 | Safety | -FHL | 21 |
| 5. | CON | CONVENTIONS AND DERIVATIONS | | |
| | 5.1 | 1 Definition of Baseline | | |
| | 5.2 | Definition of Day 1 | | |
| | | 5.2.1 | GL Treatment | |
| | | 5.2.2 | FHL Treatment | 22 |
| | 5.3 | Demog | graphic and Disposition | 22 |
| | 5.4 | Prior a | and Concomitant Medications | 22 |
| | 5.7 | FACE-Q | | |
| | 5.8 | Advers | se Events | 24 |
| 6. | STA | TATISTICAL METHODS | | |
| | 6.1 | Subjec | et Disposition | 24 |
| | 6.2 | 2 Demographic and Baseline Characteristics | | |
| | 6.3 | 8 Medical History | | |
| | 6.4 | Prior and Concomitant Medications | | |
| | 6.5 | 5 Efficacy Analyses | | |
| | | 6.5.1 | Primary Efficacy Analysis | 25 |
| | | 6.5.4 | Adjustments for Covariates | 27 |
| | 6.6 | Safety | Analyses | 27 |
| | | 6.6.1 | Extent of Exposure | 27 |
| | | 6.6.2 | Injection Site Evaluations | 28 |
| | | 6.6.3 | Adverse Events | 28 |
| | | 6.6.4 | Laboratory Tests | 29 |



# LIST OF TABLES

| Table 3.3.4-1: Clinical Laboratory Test | ts | 19 |
|-----------------------------------------|----|----|
| | | 1 |

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Term |
|--------------|----------------------------------------------------------|
| AE | Adverse Event |
| CI | Confidence interval |
| DAXI | DaxibotulinumtoxinA |
| FASE | Facial Age Self Evaluation |
| DRC | Data Review Committee |
| FASE | Facial Age Self Evaluation |
| FHL | Forehead lines |
| GAIS | Global Aesthetic Improvement Scale |
| GL | Glabellar lines |
| IGA-FWS | Investigator Global Assessment Frown Wrinkle Severity |
| IGA-FHWS | Investigator Global Assessment Forehead Wrinkle Severity |
| IM | Intramuscular |
| MedDRA | Medical Dictionary for Drug Regulatory Affairs |
| PFWS | Patient Frown Wrinkle Severity |
| PFHWS | Patient Forehead Wrinkle Severity |
| PI | Principal Investigator |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| TEAE | Treatment-emergent adverse event |
| UPT | Urine pregnancy test |
| WOCBP | Women of childbearing potential |

#### 1. INTRODUCTION

The efficacy and safety of botulinum toxin type A for the treatment of FHL has been evaluated in a number of studies. Solish et al. (2016) conducted the first large-scale, multicenter study of onabotulinumtoxinA with 40 U or 30 U total injected into both the frontalis and the glabellar complex. Complementary treatment of the glabellar complex in conjunction with the frontalis provides more satisfactory results and reduces the potential for eyebrow ptosis. At 4 weeks after the first injection, 94.4% of subjects at the 40 U dose and 84.2% of subjects at the 30 U dose were satisfied or very satisfied with the reduction in FHL severity. A longer duration of effect was noted in the 40 U dose group. There was no observed dose response noted in the incidence of eyebrow- or eyelid-related AEs in either the 40 U and 30 U dose groups. The overall incidence of eyebrow ptosis across both doses (coded as facial paresis) was low at 2.3%.



This statistical analysis plan (SAP) describes the objectives of the study and the safety and efficacy assessments that are collected. The safety endpoints and the efficacy endpoints are defined, and the statistical methods used to analyze them are presented. Table shells for the planned end-of-text tables, figures, and listings are included in a separate document, but the titles are specified following the text of the SAP.

#### 2. STUDY OBJECTIVES

## 2.1 Objectives

# 2.1.1 Primary Objective

The primary study objective is to evaluate the efficacy and safety of DaxibotulinumtoxinA (DAXI) for Injection in the treatment of dynamic Forehead Lines (Frontalis) (FHL).

# 2.2 Trial Endpoints

# 2.2.1 Efficacy Endpoints

The primary efficacy endpoint is the proportion of subjects achieving a score of 0 or 1 (none or mild) in FHL severity at maximum eyebrow elevation at 4 weeks after FHL treatment (Week 6) on the Investigator Global Assessment Forehead Wrinkle Severity (IGA-FHWS) scale.





# 2.2.2 Safety Endpoints

The primary safety endpoint is the incidence, severity, and relationship to study drug of TEAEs and SAEs during the overall study duration.

## 3. OVERALL STUDY DESIGN AND PLAN

## 3.1 Study Design

This is a phase 2a, multicenter, open-label, dose-escalation study to evaluate the safety and efficacy of DAXI for injection for the treatment of subjects with moderate to severe FHL in conjunction with GL treatment. This study will be conducted at 4 sites in the United States and Canada.



A Data Review Committee (DRC) will be used to review data from each cohort and will determine whether to proceed to the next cohort. If the DRC elects not to proceed with the FHL injection in a given dose cohort, subjects assigned to that cohort who have already received GL treatment will be followed for 14 weeks from the time of treatment (Day 1).









## 3.1.1 Determination of Sample Size



#### 3.1.2 Treatments Administered

This is an open-label, non-randomized study. Subjects will be sequentially enrolled by cohort. All subjects will receive DAXI for injection according to assigned cohort.

## 3.2 Efficacy and Safety Assessments

The primary efficacy assessments will include investigator assessment of GL and FHL severity and improvement on the IGA-FWS and IGA-FHWS, respectively as well as subject assessment of severity and improvement of GL and FHL on the PFWS and PFHWS, respectively.

# **3.2.1** Frown and Forehead Wrinkle Severity

Frown wrinkle severity is assessed by both the subject (PFWS) and the investigator (IGA-FWS) using the same 4-point rating scale, where scores range from 0 = none to 3 = severe.

Forehead wrinkle severity is assessed by both the subject (PFHWS) and the investigator (IGA-FHWS) using the same 4-point rating scale, where scores range from 0 = none to 3 = severe.

#### 3.2.2 Patient Global Satisfaction with Treatment

At each clinic visit after treatment, the subject will be asked to complete the Subject Global Satisfaction with Treatment Questionnaire to rate their satisfaction with the treatment results using a 7-point scale. The scale ranges from 0 = Very Dissatisfied to 6 = Very Satisfied, with a rating of 3 = Neither Satisfied nor Dissatisfied.

## 3.2.3 Global Aesthetic Improvement Scale

The Investigator and subject will assess the visual appearance (at maximum eyebrow elevation) of the improvement from the baseline condition in FHL and in visual appearance in the improvement of GL during maximum frown using the 7-point severity GAIS. The scale ranges from -3 = Very much worse to 3 = Very much improved, with a rating of 0 = No change.

# 3.2.5 Facial Age Self Evaluation

At each clinic visit, the subject will be asked to rate their perceived age using the FASE questionnaire (see Appendix 9 of the protocol).

# 3.2.6 FACE- $Q^{TM}$

At each clinic visit, the subject will be asked to complete the FACE-QTM Satisfaction with Forehead and Eyebrows and the FACE-QTM Appraisal of Lines: Forehead questionnaires (see Appendix 11 of the protocol). The questionnaires ask subjects to rate how bothered they are by their FHL using 6 questions about general appearance with a rating scale of 1 to 4 with 1 = Not Bothered and 4 = Extremely Bothered. The final question related to the number of forehead lines was not included in the study assessment.



## 3.3 Safety Assessments

#### 3.3.1 Adverse Events

All adverse events (AEs) will be recorded and classified on the basis of MedDRA terminology. AE severity will be graded as mild, moderate, or severe as defined in Section 9.3.2 of the protocol. Relationship of an AE will be graded as definite, probable, possible, or unrelated. AEs with an onset on or after the date and time of trial treatment or events which were present before treatment and which worsened after treatment will be considered as treatment-emergent.

AEs with missing severity will be considered as "severe". AEs with missing relationship will be considered as "related". If the start of an AE relative to the administration of trial treatment cannot be definitively determined, it will be considered to have occurred after treatment and the event considered as treatment-emergent.



## 3.3.3 Injection Site Evaluation

Injection sites will be evaluated at screening for signs of skin inflammation or active disease. The GL treatment areas will be evaluated at Day 1 (pre- and post-treatment) and at Weeks 2 and 4. The FHL treatment areas will be evaluated at Week 2 (pre- and post-treatment) and at Weeks 4 and 6. The

assessment will be done as a global evaluation of the 5 injection sites for GL and 3 injection sites for FHL. The presence of erythema, edema, burning or stinging, itching or bruising will be captured as medical history (pre-treatment) or as an AE (post-treatment).

## 3.3.4 Clinical Laboratory Data

As outlined in Table 3.3.4-1, non-fasting samples for hematology, chemistry, PT (screening only) and urinalysis will be collected at screening, the Week 4 Visit, and the Week 38 or Final Evaluation Visit.

Urinalysis will be evaluated at the study center.

Urine pregnancy tests (UPT) will be performed at screening, prior to treatment administration at Baseline and Week 2, and at the Week 38 or Final Evaluation Visit. A serum pregnancy test will be performed to confirm pregnancy whenever a post-treatment UPT is positive.

**Table 3.3.4-1: Clinical Laboratory Tests** 

| <b>Serum Chemistry</b> | Hematology | Urinalysis | Additional Tests |
|---|---|---|---|
| Glucose | Hemoglobin | Specific gravity | Prothrombin time (PT) (screening only) |
| Total bilirubin | Hematocrit | pН | |
| Alanine | Leukocyte Count (total) | Glucose | UPT (WOCBP only)* |
| aminotransferase | | Protein | |
| Aspartate | Leukocyte Count (differential) | Blood | |
| aminotransferase | | Bilirubin | |
| Alkaline phosphatase | Red Blood Cell<br>Count | Ketones | |
| Blood urea nitrogen | Platelet Count | | |

WOCBP = Women of child-bearing potential



## 3.3.6 Vital Signs

Vital signs (i.e., body temperature, respiration rate, sitting radial pulse rate, and sitting systolic and diastolic blood pressures) will be obtained at the screening, Day 1, Week 2, and Week 38 or Final Evaluation Visits,

New abnormal findings or worsening from baseline (Day 1 prior to GL treatment) at subsequent assessments, if judged clinically significant, should be recorded as an AE.

## 3.3.7 Physical Examination

A targeted physical examination, will be conducted at screening, Day 1, Week 2 and Final Evaluation Visits. Significant physical examination findings that are present prior to investigational product administration will be reported as Medical History.

Significant physical examination findings after investigational product administration which meet the definition of an AE will be recorded as an AE.



## 3.4 Interim Analyses and Data Monitoring

#### 3.4.1 Data Review Committee

Due to the dose-escalation nature of the study design, safety data and subject photographs/videos will be evaluated by the DRC at Week 5 following GL treatment (3 weeks after FHL treatment) for each cohort before a decision is made to move forward with the next and subsequent doses. If the DRC elects not to

proceed with the FHL injection in a given dose cohort, subjects will be followed for 14 weeks from the time of treatment (Day 1).

Dose escalation for FHL may be stopped at the discretion of the DRC as outlined in the DRC Charter. The full details for the roles and responsibilities of the DRC will be detailed in the study-specific DRC charter.

## 3.4.2 Interim Analysis

A formal interim analysis of the data will be performed when all subjects finish 8 weeks after receiving the FHL treatment or have withdrawn from the study earlier. This interim analysis will be a high level analysis of study conduct, efficacy and safety. The analysis will be performed by the study team in a restricted access folder. Efficacy will focus on the primary and secondary endpoints.

Individual tables, listings, and figures to be included in the interim analyses are denoted in Section 9 below with an asterisk.

#### 4. ANALYSIS POPULATIONS AND SUMMARY GROUPS

Five analysis populations will be specified, ignoring cohort membership. These populations are: Enrolled, GL-Evaluable, FHL-Evaluable, Safety and Safety-FHL. Analyses performed on the Enrolled, GL-Evaluable and FHL-Evaluable population will utilize the planned treatment assignment(s). Analyses performed on the Safety and Safety-FHL populations will utilize the actual treatment(s) received.

## 4.1 Enrolled Population

All subjects who receive the GL treatment. A subject will be considered "enrolled" if they receive any investigational product including a partial dose.

## 4.2 GL-Evaluable Population

All enrolled subjects who have any post-GL treatment assessment of IGA-FWS at maximum frown.

# 4.3 FHL-Evaluable Population

All enrolled subjects who receive the FHL treatment and have any post-FHL treatment assessment of IGA-FHWS at maximum eyebrow elevation.

## 4.4 Safety Population

All enrolled subjects.

## 4.5 Safety-FHL

All enrolled subjects who receive the FHL treatment.



Cohort 4: DAXI 30 U

#### 5. CONVENTIONS AND DERIVATIONS

#### **5.1** Definition of Baseline

The baseline value will be the last available non-missing value prior to GL treatment on Day 1. Assessments taken on the same day as GL treatment will be assumed to be prior to treatment unless indicated to be obtained post-treatment.

## 5.2 Definition of Day 1

#### **5.2.1 GL** Treatment

Study Day 1 is defined as the day of the DAXI 40 U dose for GL treatment. All time-to-event analyses for assessments of GL will utilize the date of study day 1 as the start date.

#### **5.2.2 FHL Treatment**

Day 1 of FHL treatment is defined as the day of DAXI dose for FHL treatment. All time-to-event analyses for assessments of FHL will utilize the date of FHL treatment as the start date.

Note that this definition allows for delays in administration of DAXI for FHL treatment and requires a relative day variable to be derived for days post-FHL treatment.

## 5.3 Demographic and Disposition

Age in years at time of enrollment will be derived relative to the date of informed consent as (consent date – date of birth + 1)/365.25 and truncated to 0 decimal points. Age will also be categorized into two groups: <65 years and  $\ge65$  years.

## **5.4** Prior and Concomitant Medications

Prior therapies and medications are those which began and were stopped before receipt of study medication. Concomitant therapies and medications are those which were ongoing at the receipt of study medication and those which were taken during the study (i.e., between the date of first dose and the last study visit).



## 5.7 FACE-Q

The FACE-Q assessments will be scored and converted to a transformed score which ranges from 0 to 100 according to scoring rules for the assessment. Section 8.1 for scoring of the FACE-Q Satisfaction with Forehead and Eyebrows; and, Section 8.2 for scoring of the FACE-Q Appraisal of Lines: Forehead.

#### 5.8 Adverse Events

Treatment-emergent AEs are those AEs with an onset on or after the date and time of trial treatment or events which were present before treatment and which worsened after treatment.

AEs with missing severity will be summarized as "severe". AEs with missing relationship will be summarized as "related".

#### 6. STATISTICAL METHODS

All statistical programming will be performed using statistical analysis system (SAS) version 9.4 or higher.



#### 6.1 Subject Disposition

The number and percentage of subjects who have signed informed consent, enrolled, received each treatment (GL and FHL), and completed visits will be tabulated by summary cohort and overall; and, included in a listing. Reasons for not completing the study will also be tabulated by summary cohort and overall using numbers and percentages; this data will also be included in a listing. For those subjects who are considered to have failed screening, the reason(s) for failure will be provided in a listing.

The number and percentage of subjects included and excluded from the analysis populations will be tabulated overall and for each summary cohort. Reason(s) for exclusion from each population will be summarized and listed.

A summary of the duration of the subject participation in the study will be produced, including the n, mean, standard deviation (SD), median, first and third quartiles, minimum, and maximum duration in weeks, as well as the number and percentage of subjects in the duration categories.

Major protocol deviations will be listed and summarized by summary group.

## 6.2 Demographic and Baseline Characteristics

Descriptive statistics will be used to summarize demographic and baseline characteristics by summary cohort and overall.

Demographic data include age, age category, sex, ethnicity, and race. Baseline characteristics include prior Botulinum toxin Type in the GL and FHL, time since last prior Botulinum toxin Type A injection in the GL and FHL, and Fitzpatrick skin type, as well as the baseline values of the efficacy assessments, PFWS, PHFWS, IGA-FWS, and IGA-FHWS. Summaries will be produced for the Enrolled population. If the GL Evaluable, FHL Evaluable, or Safety FHL population differs from the Enrolled population, then the summaries will be produced for the population(s) which differ from the Enrolled population.

## 6.3 Medical History

Medical history will be classified on the basis of MedDRA terminology, using the latest terminology at the time of database finalization. Medical history will be summarized for the Safety FHL population by summary cohort and overall, by system organ class, and by preferred term; and, will be listed.

## 6.4 Prior and Concomitant Medications

Prior therapies/medications and concomitant therapies/medications will be coded using the World Health Organization (WHO) drug dictionary and summarized by Anatomical Therapeutic Chemical (ATC) second level term and Preferred Name for the Safety population. Prior and concomitant medications will be summarized separately.

# 6.5 Efficacy Analyses

Descriptive statistics will be provided for all efficacy variables at all visits by cohort. A 95% exact CI will be provided for proportions. All analyses displaying proportions will use population counts as denominators at all visits regardless of the number of actual observations recorded. Differences between cohorts will not be presented except where specifically identified in the shells.

The Efficacy GL population will be used when analyzing endpoints associated with GL.

The Efficacy FHL population will be used when analyzing endpoints associated with FHL.

## 6.5.1 Primary Efficacy Analysis

The proportion of subjects achieving a score of 0 or 1 (none or mild) on the IGA-FHWS at maximum eyebrow elevation at Week 6 will be summarized. Subjects with no data at Week 6 after imputation of worst value will be considered to not meet the criteria (i.e., are imputed as non-responders). An exact 95% confidence intervals for the individual proportions will also be provided. A Cochran-Mantel-Haenszel test of association, stratified by stratified by baseline IGA-FHWS severity and study center, will be performed. In addition, an exact Cochran-Armitage test for trend, ignoring the stratification factors, will be performed. If the Cochram-Mantel-Haenszel test is significant at the 0.05 significance

level, then a linear regression on response will be performed with categorical dose as the predictor. An unstratified logistic regression analysis may still be used to explore the dose-response relationship.



# 6.5.3.1 Proportions of Subjects Meeting a Given Criterion

The assessments of the proportion of subjects meeting a given criterion ("responders") will be summarized by summary cohort and visit. For each endpoint at selected visits, the point estimates and exact 95% CIs will be computed using the same methods as with the primary endpoint.

The proportion of responders will also be graphically displayed in a plot with time on the x-axis and the proportion of subjects responding on the y-axis.

## 6.5.3.2 Time to Return to, or Time to Loss of, a Given State

The time to return to a given state, or time to loss of a given criterion, will be summarized with point estimates of median duration and 2-sided, 95% CIs, using the log-log transformation by summary cohort. Estimates of survival rates and the 2-sided, 95% CI, using the log-log transformation will also be provided. Kaplan-Meier survival curves will be plotted such that each summary group is a separate line in the same plot.



# 6.5.3.4 Descriptive Statistics and Change from Baseline

Responses to the FASE questionnaire at the Week 2 study visit, actual age, number of years older, younger will be descriptively summarized.

Transformed scores for the FACE-Q<sup>TM</sup> Satisfaction with Forehead and Eyebrows and the FACE-Q<sup>TM</sup> Appraisal of Lines: Forehead will be summarized using descriptive statistics for continuous variables.

## 6.5.4 Adjustments for Covariates

The analysis of the primary endpoint requires a stratified exact logistic regression model be run, where the strata are created based on the baseline IGA-FHWS severity and study site, both of which are considered to be covariates.



## 6.6 Safety Analyses

Safety summaries and analyses will be performed on the Safety and Safety FHL populations and will be presented by cohort and in total across cohorts. Descriptive statistics will be presented to summarize the safety data. By visit safety summaries will use denominators based on the number of subjects with valid observations at that visit unless otherwise specified.

# 6.6.1 Extent of Exposure

All subjects are planned to receive two treatments of investigational product (GL, FHL treatments). The dosage of investigational product injected and the dose of investigational product injected at each of the injection sites will be summarized overall and by summary cohort for each administration using

descriptive statistics (number of non-missing observations, mean, median, first and third quartiles, minimum, maximum, and standard deviation).

## **6.6.2** Injection Site Evaluations

The injection site evaluations for GL and FHL will be summarized separately using number and percentage of subjects with a reaction at any post-treatment visit. In addition, the number and percentage of subjects experiencing an AE of special interest related to GL injection site reactions and FHL injection site reactions will be summarized by summary cohort, system organ class, and preferred term.

#### 6.6.3 Adverse Events

All AEs will be recorded and classified on the basis of MedDRA terminology. All treatment-emergent AEs will be summarized by summary cohort and overall, system organ class, preferred term, severity, and seriousness. When summarizing events by causality and severity by subject, each subject will be counted only once within a system organ class or a preferred term by using the event with the greatest relationship and highest severity within each classification. Additionally, some summaries will present the number of AEs as well as incidence.

An overall summary of treatment-emergent AEs (TEAEs) will be provided. The number and percentage of subjects experiencing an AE, an SAE, a related AE, a related SAE, an AE of special interest, an AE leading to study discontinuation, and an AE resulting in death will be summarized.



All information pertaining to AEs noted during the trial will be listed by subject, detailing the verbatim description given by the Investigator, preferred term, system organ class, start date, stop date, severity, action taken regarding trial drug, corrective treatment, outcome, and drug relatedness. The event onset relative (in number of days) to the date of treatment for GL and FHL, as well as to the date of last treatment administration prior to the event, will be provided. In addition, a list of adverse events that lead to the subject's premature discontinuation of the trial will be provided. Serious adverse events (SAEs) will be listed by subject.

## 6.6.4 Laboratory Tests

## 6.6.4.1 Clinical Safety Laboratory Parameters

Laboratory test results will be summarized with descriptive statistics by visit. Change from baseline to post-baseline visits will be summarized for continuous test results. A summary of abnormal urinalysis incidence will be presented displaying normal, abnormal (not clinically significant), and abnormal (clinically significant) results.

Shift tables will be presented to summarize laboratory test results at Baseline and Final Evaluation Visit. Normal ranges established by the central laboratory will be used to determine shifts. A listing of all out-of-range laboratory test results at any evaluation will also be provided. Determination of clinical significance for all out-of-range laboratory values will be made by the investigator and included in the listing. In addition, a listing of all clinically significant laboratory test results will be provided.

# 6.6.4.2 Pregnancy Tests

Urine pregnancy tests will be presented in data listings for all treated subjects in the category of woman of child-bearing potential.



## 6.6.6 Vital Signs and Physical Examination

Vital signs and ECG parameters will be summarized by cohort with descriptive statistics by visit. Vital signs and ECG parameters will summarize the actual value as well as the change from baseline for each visit for continuous parameters.

Abnormal findings from the physical examination will be summarized by body system and cohort using number and percentage of subjects with a normal, abnormal and clinically significant, or abnormal and not clinically significant result.

## 6.7 Changes from the Planned Analyses

The primary analysis to explore dose response was planned to be an exact logistic regression stratified by study center and baseline severity, however, the conditional distribution is degenerate. A logistic regression may still be performed, but the primary analysis has been changed to a Cochran-Mantel-Haenszel statistic supplemented with the Cochran-Armitage test for trend. If the Cochran-Mantel-Haenszel test is significant, then a linear regression with dose as the predictor will be performed.





